CLINICAL TRIAL: NCT07002866
Title: Suubi4PrEP: Improving PrEP Access and Adherence Among Adolescent Girls and Young Women in Uganda
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Makerere University (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Fred Ssewamala, William E. Gordon Distinguished Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH139471 (NIH)
Record Dates: First submitted 2025-05-17; First posted 2025-06-04 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: HIV Prevention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm: Bolstered Treatment (Experimental): Participants in this arm will receive 5 sessions of HIV risk reduction (HIVRR) that incorporates sessions on PrEP, aimed at strengthening HIV prevention, knowledge and skills. Sessions will be delivered by trained community healthcare workers.
  Interventions: Behavioral: HIV Risk Reduction (HIVRR)
- Treatment arm I: HIVRR+PS (Experimental): Participants randomized to this arm will receive 5 sessions of HIVRR (described about) and will engage with PrEP peer supporters (PS). Peers will be women currently on PrEP willing to share their lived experiences. Women will meet with peer supporters at least 8 times during the intervention period. Meetings will last approximately 1-hour and will explore the cost-benefits of service utilization and to problem solve how to overcome individual barriers to PrEP access, utilization and adherence.
  Interventions: Behavioral: HIV Risk Reduction (HIVRR); Behavioral: PrEP Peer Supporters (PS)
- Treatment arm II: HIVRR+PS+EE (Experimental): The economic empowerment (EE) intervention will be in the form of a matched savings account (MSA) plus financial literacy (FL) sessions. Participants enrolled in the combination intervention arm will receive 5 sessions of HIVRR and PrEP peer supporters (as described above) and a MSA. Specifically, our partnering banks will open up matched savings accounts for the participants in their name. Participants will save money in their matched savings accounts over a 20-month period. The study team will monitor the accounts using the statements received directly from the banks holding the accounts. Participants will receive monthly bank statements indicating their own savings and the associated match (1:1 match rate). They will also receive eight financial literacy (FL) sessions.
  Interventions: Behavioral: HIV Risk Reduction (HIVRR); Behavioral: PrEP Peer Supporters (PS); Behavioral: Matched Savings Accounts + Financial Literacy (FL)

INTERVENTIONS:
Behavioral: HIV Risk Reduction (HIVRR) — This is an intervention comprised of 5 sessions of an evidence-based, HIV/STI risk reduction with PrEP to strengthen HIV prevention knowledge and behavioral skills intervention. Session content cover harm reduction, social support networks, HIV knowledge, transmission risks and testing procedures for HIV/STIs, build enthusiasm for condom use, alternatives to unsafe sex, importance of safer sex negotiations, strategies to negotiate safer sex, setting appropriate risk reduction goals, introduction to PrEP, PrEP screening and eligibility; monitoring and managing PrEP side effects and stigma, recognizing and understanding consequences of abusive behavior by any sexual partners or others; build safety plan skills; review and identify ways to increase social support; build skill in communication with health care professionals.
Behavioral: PrEP Peer Supporters (PS) — PrEP peer supporter are women currently on PrEP willing to share their lived experiences. Women will meet with peer supporters in a group at least 8 times during the intervention period (every 2-3 months). Sessions with peers will involve unstructured, in-depth discussions that integrate peers' own lived experiences and emerging PrEP-related issues as raised by participants. These may include, how to mitigate PrEP stigma and disclosure, creating PrEP adherence strategies, navigating family and intimate relationship issues, and navigating provider attitudes. At each stage of the facility visit (waiting space, consultation, and pharmacy), peer supporters will explain facility protocols, and strategies women can use to overcome facility-level barriers to care.
  Arms: Treatment arm I: HIVRR+PS; Treatment arm II: HIVRR+PS+EE
Behavioral: Matched Savings Accounts + Financial Literacy (FL) — A matched savings account (MSA) is a savings account held at a local bank whereby deposits made by the participants are matched by the intervention to encourage savings and investment in skills and asset development. The accounts introduce participants to financial management skills, introduce them to formal financial institutions, and by matching their deposits, incentivize women to save small amounts. Each participant will receive an account held in her own name, and will be allowed to save an equivalent of US$10 a month or US$200 for the 20-months intervention period. During the intervention period, participants will have direct access to both their personal savings deposited in the accounts and the match provided by the study. In addition, participants will also receive six 1-2-hour financial literacy (FL) workshop sessions that cover components on saving, and financial management.
  Arms: Treatment arm II: HIVRR+PS+EE

SUMMARY:
The study will employ a multilevel combination intervention focused on PrEP initiation and adherence among adolescent girls and young women (AGYW) (aged 15-24) living in HIV hotpots in Uganda. Specifically, the study will combine: 1) HIV risk reduction (HIVRR) that incorporates sessions on PrEP, 2) Peer Supporters (PS) with lived experiences taking PrEP to facilitate linkage to and continued care, share strategies to address misconceptions, manage disclosure and stigma, and model positive lifestyles while engaging in care services, and 3) an economic empowerment (EE) component that includes a matched savings account and financial literacy targeting poverty and financial barriers associated with PrEP access. Working within 30 health care systems, we will randomly assign 600 AGYW (at the community level) to one of three study arms (n=200 AGYW, n=10 sites per arm): 1) HIVRR only, 2) HIVRR+ PS, or 3) HIVRR + PS + EE. The interventions will be implemented for 20 months, and data collected at baseline, 12, 24, 36 months.

DETAILED DESCRIPTION:
Adolescent girls and young women (AGYW) aged 15-24 are twice as likely to be living with HIV than young men in Sub-Saharan Africa (SSA). HIV prevention strategies available to AGYW primarily depend on male partner cooperation, limiting the ability for these strategies to reduce HIV spread. Oral pre-exposure prophylaxis (PrEP) is a highly effective biomedical HIV prevention method. However, as effective as PrEP has been, it is underutilized. Lack of social support, disclosure concerns, stigma and discrimination, financial costs associated with transport to clinics and food to accompany medication are still major barriers. Peer support interventions and PrEP awareness via peers has been associated with increased PrEP uptake. However, these approaches may not be as effective when delivered alone -given that poverty-associated factors, too, greatly undermine PrEP access, uptake and adherence. Thus, combining multilevel interventions, in this case, combining peer support with economic empowerment (EE) targeting poverty and financial constraints, may offer additive effects to overcome these barriers. We propose a multilevel combination intervention focused on PrEP initiation and adherence among AGYW living in HIV hotpots in Uganda. Suubi(hope)4PrEP will combine: 1) HIVRR that incorporates sessions on PrEP, 2) peer supporters (PS) with lived experiences taking PrEP to facilitate linkage to and continued care, and 3) EE components targeting financial barriers associated with PrEP access. We will randomly assign 600 AGYW (at the community level) to one of the three study arms (n=200 AGYW, n=10 sites per arm): 1) HIVRR only, 2) HIVRR+ PS, or 3) HIVRR + PS + EE. Specific aims are:

Aim 1. Examine the impact of Suubi4PrEP on PrEP initiation and adherence.

Aim 2. Examine the effect of Suubi4PrEP on hypothesized mechanisms of change and intervention mediation.

Aim 3. Use mixed methods to explore multi-level factors that influence PrEP initiation and adherence.

Aim 4. Assess the cost and cost-effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-24 years
2. At a high risk of HIV. AGYW will be deemed to be at substantial risk, and eligible to participate in the study, if they report at least one of the seven high-risk sexual behaviors on the risk assessment tool: 1) vaginal/anal sexual intercourse with more than one partner of unknown HIV status in the past six months, 2) vaginal/anal sex without a condom in the past six months, 3) sex in exchange for money, goods or a service in the last six months, 4) injecting drugs in the past six months, 5) diagnosis with an STI more than once in the past twelve months, 6) post-exposure prophylaxis (PEP) for sexual exposure to HIV in the past six months, and 7) having an HIV-infected sexual partner who was not on ART.

Exclusion Criteria:

1. HIV positive
2. Unable to understand the study procedures and/or participant rights during the informed consent process
3. Unwilling or unable to commit to completing the study

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants must be female
Enrollment: 600 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
PrEP Initiation | Baseline, 12, 24 and 36 months
  Proportion of eligible participants who initiate PrEP

SECONDARY OUTCOMES:
PrEP Adherence | Baseline, 12, 24, 36 months
  PrEP adherence will be assessed using biological data (Tenofovir drug levels in urine). High urine tenofovir levels indicate good adherence to PrEP medication, while low or undetectable urine tenofovir levels indicate non-adherence to PrEP.

CONTACTS AND LOCATIONS:
Locations (2):
- Washington University in St. Louis, St Louis, Missouri, United States
- International Center for Child Health and Development (ICHAD), Masaka, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Once all of the data has been de-identified, cleaned, and validated, and main findings have been published, the Investigators expect to share data with the scientific community. The research team will make datasets available to any individual who makes a direct request to the PIs and indicates the data will be used for the purposes of research (per CFR Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge."). In sharing participant data, the team will follow Brown School of Social Work Office of Sponsored Projects' data sharing agreements.